CLINICAL TRIAL: NCT02455336
Title: An Open Label Safety and Efficacy Trial of Fenofibrate in Persons With SCI
Brief Title: Fenofibrate Treatment in SCI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1925-P
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injury; Dyslipidemia
Keywords: tetraplegia; paraplegia; hypertriglyceridemia; hyperlipidemia; peroxisome proliferator-activated receptor alpha
MeSH Terms: conditions — Spinal Cord Injuries; Dyslipidemias; Quadriplegia; Paraplegia; Hypertriglyceridemia; Hyperlipidemias | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fenofibrate (Experimental): Subjects with adverse TG concentrations (i.e., paraplegia: >/=135 mg/dl; tetraplegia >/=115 mg/dl) will be randomized to receive once daily fenofibrate therapy (i.e., 145 mg) for 4 months
  Interventions: Drug: Fenofibrate
- No Intervention (Other): Subjects with adverse TG concentrations (i.e., paraplegia: >/=135 mg/dl; tetraplegia >/=115 mg/dl) will be randomized to receive no therapy for 4 months
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate is a peroxisome proliferator-activated receptor alpha agonist that is demonstrated to reduce triglyceride concentrations in the blood.
  Arms: Fenofibrate
Other: No intervention — A cohort of participants will be randomized to receive no study drug, but will engage in study encounters.
  Arms: No Intervention

SUMMARY:
Cardiovascular disease-related morbidity in persons with spinal cord injury (SCI) occurs earlier in life, at a greater prevalence than that of the general population, and is the primary cause of death after the first year of injury. During the chronic phase of SCI, a characteristic dyslipidemia emerges, which is characterized by low serum high density lipoprotein cholesterol (HDL-C) concentrations, with values often qualifying to be an independent risk factor for coronary artery disease, and elevations in serum triglycerides (TG). Serum low density lipoprotein cholesterol concentrations in those with SCI are usually similar to those of the general population. The current proposal in persons with SCI aims to determine the safety and efficacy of short-term fenofibrate treatment, an anti-lipid medication whose primary action lowers serum TG and raises serum HDL-C levels.

DETAILED DESCRIPTION:
Although considered a modifiable risk factor for coronary artery disease (CAD) in the general population, the magnitude of physical activity required to promote cardiorespiratory fitness and a clinically meaningful change in blood-derived biomarkers of CAD is not achievable in those with a severe physical disability, such as with immobilizing paralysis from spinal cord injury (SCI). During the chronic phase of SCI, a characteristic dyslipidemia emerges, with mean serum high density lipoprotein cholesterol (HDL-C) concentrations <40 mg/dl, a threshold level for HDL-C that is appreciated to be an independent risk factor for CAD, elevations in triglycerides (TG) to concentrations at, or near, target values for the general population that trigger clinical intervention, and low density lipoprotein cholesterol (LDL-C) concentrations that are within the normal range. It should not be a surprise that cardiovascular disease (CVD)-related morbidity in persons with SCI occurs earlier in life, at a greater prevalence than that of the general population, and is the primary cause of death after the first year of injury. Population-based epidemiological studies are unavailable for clinical guidance because of the relatively low incidence rates for SCI. Clinical target values used to initiate treatment in the general population may be inappropriate in those with SCI because of their unique pathophysiology. In the absence of significant physical activity and lifestyle modifications, it would seem that appropriate pharmaceutical options are needed to properly manage markers of CVD-related risk in persons with SCI. To date, there is limited empirical evidence to support the use of lipid-lowering treatments in persons with SCI.

Fenofibrate is a fibric acid derivate that activates peroxisome proliferator-activated receptor and lipoprotein lipase, leading to enhanced elimination of TG from plasma. In clinical trials where fenofibrate was used as a monotherapy, serum TG concentrations fell 41-53%, very low density lipoprotein (VLDL) fell 38-52%, LDL-C decreased 6-20%, and HDL-C improved by as much as 20%. In consideration for the nature of dyslipidemia in persons with SCI, fenofibrate appears to be an appropriate first-line agent for treatment in this cohort, especially because most of those with SCI have LDL values that are within the clinically acceptable range. In the general population, standard clinical practice for lipid-lowering treatment with fenofibrate monotherapy follows a known and clinically accepted timeline to monitor safety and to determine therapeutic efficacy. It is recommended that, if after 2 months of continuous therapy there are no beneficial changes to the lipoprotein profile, that treatment be discontinued (i.e., non-responders). Similarly, several large clinical trials have demonstrated that the peak therapeutic effects of fenofibrate are observed after 12-16 weeks of treatment (i.e., responders). The proposed study will test the efficacy of administering fenofibrate to persons with SCI, a severely immobilized cohort that does not have established clinical practice guidelines to treat dyslipidemia and appears to have unique considerations that may be hypothesized to call for a more disease-specific approach for care. If successful, the treatment will reduce clinical markers of CVD-related risk by modifying the concentration and number of particles that are known to contribute to incident cardiac events and mortality. It is anticipated that the insight gained from this investigation will provide clinicians with a proof-of-concept for instituting appropriate use of lipid lowering agents to treat the dyslipidemia that has been well described in persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 21 to 69;
* Chronic (e.g., duration of injury at least 6 months), stable SCI (regardless of level of neurological lesion);
* American Spinal Injury Association Impairment Scale (AIS) designation of A, B or C; and
* TG concentration 135 mg/dl (paraplegia) or 115 mg/dl (tetraplegia).

Exclusion Criteria:

* Acute illness or infection;
* Reduced kidney function (by glomerular filtration rate (GFR <60 ml/min) or liver function tests (LFTs 2.5 standard deviations above the upper limit of normal);
* Current pharmacological treatment with: HMG-CoA reductase inhibitors (statins), or any other hypolipidemic agent; anti-coagulant therapy; cyclosporine; or any other medications known to effect the TG concentration (i.e., -blockers, thiazides or estrogen);
* Hypersensitivity to fenofibrate;
* Existing diagnosis of atherosclerosis, congestive heart failure, or recent history of myocardial infarction (i.e., 12 months);
* Pregnancy or women who may become pregnant during the course of the study, or those who are nursing;
* Diminished mental capacity; and
* Inability or unwillingness of subject to provide informed consent.
* Existing diagnosis of diabetes mellitus, or the results from screening blood tests indicate that diabetes mellitus is present (and perhaps undiagnosed); laboratory thresholds for exclusion will be as follows: HbA1C 6.5% and fasting plasma glucose is >126 mg/dl.

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F LaFountaine, EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fenofibrate | No Intervention
Started | 15 | 8
Completed | 10 | 6
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Non-responder to treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: Only those participants who completed the 4 month trial are included in the analysis. Three participants who experienced adverse events that discontinued the trial do not appear in the results. Two participants who did not respond to 2 months of treatment do not appear in the results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate | No Intervention | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 44 (13) | 46 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Triglyceride Concentration (Percent Change From Baseline)
Description: To determine the efficacy of fenofibrate monotherapy after 2 months of treatment to improve the lipoprotein profile; a successful response will be defined as a 25% reduction in the serum TG concentration at 2 months.
Time Frame: two months from initiating drug treatment
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Fenofibrate | No Intervention
Number analyzed (Participants) | 10 | 8
percent change from baseline | -40 (12) | -2 (16)

2. Secondary Outcome: Triglyceride Concentration (Percent Change From Baseline)
Description: To determine the efficacy of fenofibrate monotherapy to lower TG concentration at 4 months of treatment, when the peak therapeutic efficacy to drug treatment has been reported to occur.
Time Frame: four months from initiating drug treatment
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Fenofibrate | No Intervention
Number analyzed (Participants) | 10 | 8
percent change from baseline | -40 (20) | 7 (14)

3. Other Pre Specified Outcome: Adverse Event Profile
Description: Documentation and description of adverse events will be obtained in subjects who have received drug treatment compared to events occurring in the control group.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate | No Intervention
Number analyzed (Participants) | 15 | 8
Participants
  Elevated liver enzymes | 2 | 0
  Gastrointestinal discomfort | 2 | 0

ADVERSE EVENTS:
Time Frame: All blood sample results were reviewed by the study physician for the presence of adverse findings at each monthly visit during the 4 months of the treatment trial.
Description: The presence of an adverse finding in liver function tests, kidney function, CBC w/diff, or a change in the patient self-report health status were submitted to the Institutional Review Board (IRB) as an adverse event; the nature/severity of the event may have resulted in discontinuation of the subject from the study drug and continued participation in the trial, which was contingent upon the judgement of the study physician and the advice of the IRB.
Groups:
- Fenofibrate: Twenty subjects with adverse TG concentrations (i.e., paraplegia: >/=135 mg/dl; tetraplegia >/=115 mg/dl) will be randomized to receive once daily fenofibrate therapy (i.e., 145 mg) for 4 months
  Fenofibrate: Fenofibrate is a peroxisome proliferator-activated receptor alpha agonist that is demonstrated to reduce triglyceride concentrations in the blood.
- No Intervention: Ten subjects with adverse TG concentrations (i.e., paraplegia: >/=135 mg/dl; tetraplegia >/=115 mg/dl) will be randomized to receive no therapy for 4 months
  No intervention: A cohort of participants will be randomized to receive no study drug, but will engage in study encounters.
Arm/Group | Fenofibrate | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 2/15 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate (N=15) | No Intervention (N=8)
Elevated liver enzymes (Hepatobiliary disorders) | 2 (2) | 0 (0) — Elevated liver function tests (LFTs) in excess of the exclusion criterion (e.g. ≥2.5 times greater than the upper limit of normal).
Gastrointestinal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) — Experience of gastrointestinal (GI) discomfort including constipation or a change in the consistency of the stool that began shortly after initiating drug treatment or after a few weeks of use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT02455336/Prot_SAP_000.pdf